CLINICAL TRIAL: NCT06176703
Title: Mobile Application for Self-Management of Type 2 Diabetes Mellitus: Randomized Controlled Trial
Brief Title: Mobile Application for Self-Management of Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Supasuta Wongdama, Principal Investigator, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5370
Record Dates: First submitted 2023-12-05; First posted 2023-12-20 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment with mobile application in diabetes mellitus patients (Experimental)
  Interventions: Device: mobile application
- standard treatment without mobile application in diabetes mellitus patients (No Intervention)

INTERVENTIONS:
Device: mobile application — using mobile application along with standard treatment of diabetes mellitus
  Arms: Standard treatment with mobile application in diabetes mellitus patients

SUMMARY:
The goal of this Randomized Controlled Trial is to study the effect of mobile Application on glycemic control of type2 diabetes mellitus. The main questions aim to answer are:

* The effect of mobile application on glycemic control and quality of life of diabetes mellitus patients
* The satisfaction of mobile application of diabetes mellitus patients who used it Participants will be received education about diabetes mellitus and separated into two groups, intervention group(using mobile application) and control group(not using mobile application but also receive standard treatment of diabetes mellitus.

Researchers will compare intervention group to control group about glycemic control including HbA1c, complications of diabetes mellitus etc. and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Type2 diabetes mellitus who have HbA1c above 7%
* Can use application on smartphone
* age 18 years old or more (relatives are accept if participants have age more than 65 years old and cannot use smartphone)
* consent to participate the research

Exclusion Criteria:

* refuse to participate the research
* pregnancy
* using continuous glucose monitoring system or insulin pump
* disability in sight or hearing
* have been using the mobile application(RAMAdiabetes) in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-22 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | 3-6 months
  HbA1c
Glycemic control | 3-6 months
  Fasting blood sugar

SECONDARY OUTCOMES:
self-diabetes management | 3-6 months
  The Thai-Diabetes Management of Self-Efficacy Scale(T-DMSES), total score range from 19 to 95 points(minimum to maximum), each question has 1 to 5 points, higher scores mean better self diabetes management
Quality of life | 3-6 months
  The Thai version of the EQ-5D-5L Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chutintorn Sriphrapradang, Study Director — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, ฺBangkok, Thailand

IPD SHARING:
Plan to Share IPD: No